CLINICAL TRIAL: NCT00000803
Title: A Phase II Double-Blind Study of Delavirdine Mesylate ( U-90152 ) in Combination With Zidovudine ( AZT ) and/or Didanosine ( ddI ) Versus AZT and ddI Combination Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 261; 11238 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Delavirdine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Delavirdine mesylate
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To determine the safety and anti-HIV activity of delavirdine mesylate ( U-90152 ) in combination with zidovudine ( AZT ) and/or didanosine ( ddI ) versus AZT/ddI combination.

U-90152 has demonstrated anti-HIV activity. Since the combination of this drug with either AZT or ddI has synergistic inhibitory activity against HIV-1 in vitro, and triple therapy appears to have greater inhibitory activity against HIV-1 in vitro than dual therapy, the use of U-90152 in combination with AZT and/or ddI may improve the benefits of these drugs in persons with HIV disease.

DETAILED DESCRIPTION:
U-90152 has demonstrated anti-HIV activity. Since the combination of this drug with either AZT or ddI has synergistic inhibitory activity against HIV-1 in vitro, and triple therapy appears to have greater inhibitory activity against HIV-1 in vitro than dual therapy, the use of U-90152 in combination with AZT and/or ddI may improve the benefits of these drugs in persons with HIV disease.

Patients are randomized to receive U-90152/AZT/ddI, U-90152/AZT, U-90152/ddI, or AZT/ddI for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis for patients with CD4 count <= 200 cells/mm3.

Allowed:

* Topical antifungal agents.
* Oral ketoconazole, fluconazole, and itraconazole for candidiasis or disseminated fungal infections.
* Isoniazid, ethambutol, pyrazinamide, clofazimine, ciprofloxacin, and clarithromycin for acute or maintenance therapy for mycobacterial disease (also clarithromycin for MAC prophylaxis).
* Acute or maintenance therapy for toxoplasmosis.
* Acute or maintenance therapy with acyclovir (no more than 1000 mg/day) for herpes simplex virus infection.
* rEPO and rG-CSF.
* Antibiotics for bacterial infections (except rifampin and rifabutin).
* Antipyretics, analgesics, nonsteroidal anti-inflammatory agents, antiemetics, and methadone.

Concurrent Treatment:

Allowed for cutaneous Kaposi's sarcoma:

* Localized radiation therapy.
* Limited intralesional therapy.

Patients must have:

* HIV infection.
* CD4 count 100 - 500 cells/mm3.
* Prior cumulative monotherapy of <= 6 months (may have taken either AZT or ddI, but not both) OR no prior antiretroviral therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy (other than basal or squamous cell carcinoma of the skin, Stage 1 or 2 cervical intraepithelial neoplasia, or minimal Kaposi's sarcoma).
* Considered to be unlikely to comply with study requirements.

Concurrent Medication:

Excluded:

* Antiretroviral therapies and biologic response modifiers (except for study medications, rEPO, and rG-CSF).
* Rifampin.
* Rifabutin.
* Terfenadine.
* Astemizole.
* Loratadine.
* Quinidine.
* Digitoxin.
* Systemic corticosteroids for more than 21 consecutive days.
* Foscarnet.
* Systemic cytotoxic chemotherapy for a malignancy.

Patients with the following prior conditions are excluded:

* History of intolerance to AZT at <= 600 mg/day or ddI at <= 400 mg/day or discontinuation of either drug for toxicity.
* History of intolerance to trifluoperazine or piperazine citrate (per amendment).
* History of pancreatitis.
* History of grade 2 or worse peripheral neuropathy.
* Unexplained temperature >= 38.5 C on any 7 days within the past 30 days.
* Chronic diarrhea on any 15 days during the past 30 days.

Prior Medication:

Excluded:

* Prior foscarnet as induction or maintenance therapy.
* Prior U-90152.
* Prior ddC or d4T.
* Prior AZT/ddI in combination or taken separately at different times.
* Prior non-nucleoside reverse transcriptase inhibitors (nevirapine, atevirdine, etc.).
* Prior protease inhibitors (although patients from ACTG 282 are eligible).
* HIV-1 vaccine within the past 21 days.
* Acute treatment for a serious infection or for any opportunistic infection within the past 14 days.

Excluded within the past 30 days:

* Interferon or interleukin.
* Rifampin.
* Rifabutin.
* Terfenadine.
* Astemizole.
* Loratadine.
* Recombinant EPO or G-CSF.
* Hydroxyurea.
* SPV-30.
* Any other investigational drug.

Active drug or alcohol use.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 471
Dates: Study Completion 1997-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Friedland G, Study Chair; Fischl MA, Study Chair; Pollard R, Study Chair
Locations (32):
- United States (31):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Cornell University A2201, New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Griffit B, Morse G, Demeter L, Bassett R, Hughes M, Friedland G. Relationship between delavirdine (DLV) plasma levels, HIV RNA responses and DLV resistance during combination therapy with zidovudine (ZDV), and didanosine (ddI). Int Conf AIDS. 1998;12:52 (abstract no 12206)
- [Background] Freimuth WW, Chuang-Stein CJ, Greenwald CA, Wathen LK, Edge-Padbury BA, Cox SR, Daenzer CL, Wang Y, Carberry PA. Delavirdine (DLV) combined with zidovudine (ZDV) or didanosine (ddI) produces sustained reduction in viral burden and increases in CD4 count in early and advanced HIV-1 infection. Int Conf AIDS. 1996 Jul 7-12;11(1):22 (abstract no MoB295)
- [Background] Nokta M, Turk P. Partial restoration of HIV specific neutralizing activity (NA) of HIV infected patients receiving antiretrovial therapy: DDI/delaviridine (DLV), AZT/DLV, DDI/AZT or DDI/AZT/DLV. Int Conf AIDS. 1998;12:516 (abstract no 31108)
- [Background] Friedland GH, Pollard R, Griffith B, Hughes M, Morse G, Bassett R, Freimuth W, Demeter L, Connick E, Nevin T, Hirsch M, Fischl M. Efficacy and safety of delavirdine mesylate with zidovudine and didanosine compared with two-drug combinations of these agents in persons with HIV disease with CD4 counts of 100 to 500 cells/mm3 (ACTG 261). ACTG 261 Team. J Acquir Immune Defic Syndr. 1999 Aug 1;21(4):281-92. doi: 10.1097/00126334-199908010-00005. PMID 10428106
- [Background] Demeter LM, Meehan PM, Morse G, Gerondelis P, Dexter A, Berrios L, Cox S, Freimuth W, Reichman RC. HIV-1 drug susceptibilities and reverse transcriptase mutations in patients receiving combination therapy with didanosine and delavirdine. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Feb 1;14(2):136-44. doi: 10.1097/00042560-199702010-00006. PMID 9052722